### **Statistical Analysis Plan**

An open-label trial with TMC278 25 mg q.d. in combination with a background regimen containing 2 nucleoside/nucleotide reverse transcriptase inhibitors in HIV-1 infected subjects, who participated in TMC278 clinical trials

### Protocol TMC278-C222; Phase III

TMC278 (Rilpivirine)

Status: Approved

Date: 26 March 2018

**Prepared by:** Janssen Research and Development, a division of Janssen Pharmaceutica NV

**Document No.:** EDMS-ERI-157462123

**Compliance:** The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

#### **Confidentiality Statement**

The information in this document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by applicable law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you that is indicated as privileged or confidential.

# **TABLE OF CONTENTS**

| TABL | E OF CONTENTS | 2 |
|---|---|---|
| ABBF | REVIATIONS | ( |
| 1. | INTRODUCTION | , |
| 1.1. | Trial Objectives | |
| 1.2. | Trial Design | |
| 1.3. | Statistical Hypotheses for Trial Objectives | |
| 1.4. | Sample Size Justification | |
| 1.5. | Randomization and Blinding | |
| 1.5. | Nandomization and billiding | |
| | GENERAL ANALYSIS DEFINITIONS | 5 |
| 2.1. | Visit Windows | <del>[</del> |
| 2.1.1. | Trial Phases | <u> </u> |
| 2.1.2. | Analysis Time points | ( |
| 2.2. | Analysis Sets | |
| 2.2.1. | | |
| 3. | SUBJECT INFORMATION | 7 |
| 3.1. | Demographics and Baseline Characteristics | |
| 3.2. | Disposition Information | |
| 3.3. | Extent of Exposure | |
| 3.4. | Protocol Deviations | |
| 3. <del>4</del> .<br>3.5. | Concomitant Medications | |
| 3.6. | Adherence | |
| | EFFICACY | |
| 4.1. | Analysis Specifications | |
| 4.1.1. | | |
| 4.1.2. | | |
| 4.2. | Efficacy Endpoints | |
| 4.2.1. | CD4 <sup>+</sup> cell count | |
| 4.2.2. | Analysis Methods | 11 |
| 5. | RESISTANCE DETERMINATIONS | 11 |
| 6. | SAFETY | 4. |
| 6.1. | Adverse Events | |
| 6.2. | Clinical Laboratory Tests | |
| 6.2.1. | Overall Laboratory Safety | 12 |
| REFE | RENCES | 13 |
| A DDE | NDIY 1: ADVERSE EVENTS OF INTEREST | 1/ |
| | INIJIA I ALIVERSE EVENIS DE INTEREST | 112 |

#### **ABBREVIATIONS**

AE Adverse Event

AIDS Acquired Immunodeficiency Syndrome

ARV Antiretroviral
CI Confidence Interval
CM Concomitant medications
CRF Case Report Form

DAIDS Division of AIDS, National Institute of Allergy and Infectious Diseases, USA

DPS Data Presentation Specifications eCRF Electronic Case Report Form FDA Food and Drug Administration

HIV-1 Human immunodeficiency virus – type 1 ICH International Conference on Harmonization

ITT Intent-to-Treat

MedDRA Medical Dictionary for Regulatory Activities
NNRTI Non-Nucleoside Reverse Transcriptase Inhibitor

NRTI Nucleoside/Nucleotide Analogue Reverse Transcriptase Inhibitor

LOCF Last Observation Carried Forward

PI Protease Inhibitor
q.d. quaque die; once daily
RNA Ribonucleic acid
RPV Rilpivirine

SAE Serious Adverse Event
SAP Statistical Analysis Plan
TMC Tibotec Medicinal Compound

VF Virologic Failure

#### 1. INTRODUCTION

This statistical analysis plan (SAP) contains definitions of analysis sets, derived variables, and statistical methods for the Final analysis (Week 360) of safety and efficacy (antiviral activity) for the continued access study TMC278-C222. The data cut-off is 08 February 2018.

# 1.1. Trial Objectives

The objectives of this study were:

- <u>Primary objective</u>: to provide continued access to RPV for subjects who were randomized and treated with RPV in the Phase IIb (C204) or Phase III trials (C209 and C215).
- <u>Secondary objective</u>: to evaluate the long-term safety and tolerability of RPV 25 mg q.d. in combination with a background regimen containing 2 NRTIs. Available efficacy data will also be collected.

### 1.2. Trial Design

This was a Phase III, open label, multicenter, roll-over trial to provide continued access to RPV (rilpivirine) in HIV-1 infected subjects who were randomized and treated with RPV in the Phase IIb (C204) or Phase III trials (C209 and C215), and who continued to benefit from their ARV treatment. Information on safety and tolerability was collected. In addition, local information on viral load, ARV resistance and CD4<sup>+</sup> count was also collected.

At the baseline visit (roll-over visit), inclusion and exclusion criteria were assessed to confirm eligibility. Once eligibility criteria were met, subjects were to continue treatment with RPV 25 mg q.d. in comination with a background regimen containing 2 NRTIs.

Treatment was to be continued until one of the following criteria were met:

- Virologic failure
- Adverse event (AE)
- Pregnancy
- Loss to follow-up
- Withdrawal of consent
- Subject reached a virologic endpoint
- Sponsor's decision
- Switch to commercially available medication

Visits and assessments were to be performed based on local generally accepted standard of care (see time and events schedule in the protocol). However, it was recommended that visits be planned no less frequently than every 6 months.

Adverse event reporting was limited to:

- AEs considered a least possibly related to RPV
- AEs leading to discontinuation
- serious advese events (SAEs) and pregnancies
- Grade 3/4 rash, irrespective of causality

Other AEs were only collected if required as per local regulation.

## 1.3. Statistical Hypotheses for Trial Objectives

No formal hypothesis will be tested.

## 1.4. Sample Size Justification

No sample size calculation was done as this is a continued access single arm trial.

# 1.5. Randomization and Blinding

#### Randomization

As this was a continued access single arm trial, randomization procedures were not applicable.

### **Blinding**

Since this was an open label, continued access single-arm trial, blinding procedures were not applicable.

### 2. GENERAL ANALYSIS DEFINITIONS

### 2.1. Visit Windows

#### 2.1.1. Trial Phases

Analysis phases are constructed as follows:

 Table 1: Analysis Phases for Efficacy and Safety Analysis

| Trial phase | Start date | End date |
|---|---|---|
| Enrollment | Date of signing informed consent | Day before the start of the treatment phase. |
| Treatment | Date of the first intake<br>of RPV (in this study) | <ul> <li>If the subject died: min (date of last RPV intake + 7 days; date of death)</li> <li>Otherwise: minimum of:</li> <li>date of last RPV intake + 7 days, if missing, max(early withdrawal visit date; discontinuation date) + 7 days (early withdrawal visit date is from dataset sv and discontinuation date is dsstdtc)</li> <li>date of last contact (=dm.rfendtc which is the last complete date)</li> </ul> |
| Follow-up (not defined | End date of the | If the subject died: date of death |
| when derived End date is | Treatment phase + 1 | Otherwise: date of last contact |
| before Start date of this phase) | day | |

If the date of first intake of the study medication is missing, this should be substituted by the baseline visit date.

The number of days in the phase is defined as:

 $relday = visit \ day - reference \ day + I$  for visits on or after the reference  $relday = visit \ day - reference \ day$  for visits before the reference

where the reference day equals the actual start date of intake of RPV.

### 2.1.2. Analysis Time points

Subjects were to rollover after completion of one of the three parent trials. The baseline visit of this roll-over study coincided with the last visit of the treatment phase of the previous trial. If a subject was deemed eligible to participate in this trial, the subject was to receive trial medication at the baseline visit. After the baseline visit, subjects were to be evaluated as per local regulations, but it was advised that the duration between consecutive visits be no longer than 6 months.

All visits/assessments will be allocated to the following time points as per the table below, based on the number of days in the respective phase, calculated as "assessment date – start date of phase + 1 day" for Treatment and Follow-up phase.

The following time intervals are used for reporting of efficacy data

**Table 2:** Cut-points and Windows per 24-Week Intervals

| Phase | Target day | Analysis time point | Time interval (days) |
|-----------|------------|---------------------|----------------------|
| Treatment | 169 | Week 24 | [1, 252] |
| | 337 | Week 48 | [253, 420] |
| | 505 | Week 72 | [421, 588] |
| | 673 | Week 96 | [589, 756] |
| | 841 | Week 120 | [757, 924] |
| | 1009 | Week 144 | [925, 1092] |
| | 1177 | Week 168 | [1093, 1260] |
| | 1345 | Week192 | [1261, 1428] |
| | 1513 | Week 216 | [1429, 1596] |
| | 1681 | Week 240 | [1597, 1764] |
| | 1849 | Week 264 | [1765, 1932] |
| | 2017 | Week 288 | [1933, 2100] |
| | 2185 | Week 312 | [2101, 2268] |
| | 2353 | Week 336 | [2269, 2436] |
| | 2521 | Week 360 | $[2437, +\infty]$ |
| Follow-up | 30 | Follow-up | $[1, +\infty]$ |

Only the record prior to or on the first dose closest to target day 1 will be allocated to analysis time point 'Baseline'.

If two visits fall within the same interval, the one closest to the target day is used for the analysis displays and graphics to have only one evaluation per subject per analysis time point. However, all data are presented in the listings. If distances of both visits to the target day are equal, the visit latest in time is used.

#### **Baseline**

Baseline refers to the last visit in the parent study, which is the first visit in C222.

# 2.2. Analysis Sets

*Intent-to-treat (ITT) population*: the set of all subjects who have taken at least 1 dose of RPV, regardless of their compliance with the protocol and adherence to the dosing regimen. The intent-to-treat population will be used as primary and only population for all analyses.

### 2.2.1. Definition of Subgroups

All displays will be created by previous trial (both phase III trials, C209 and C215, will be analyzed together) and overall. The following labels will be used:

- RPV (C204)
- RPV (C209 and C215)
- All subjects

The following subgroups will be defined for **efficacy**:

- Gender
- Race
- Age (<50; >=50 to <65; >= 65 years at baseline)
- Cumulative adherence based on drug accountability (≤95%, >95%)
- Truvada in background ARV regimen (yes/no)
- Clade

The following subgroups will be defined for **Safety**:

- Truvada in ARV regimen (yes/no)
- Hepatitis B/C Co-infection (based on medical history in parent study)
- Hepatitis B infection (based on medical history in parent study)
- Hepatitis C infection (based on medical history in parent study)
- Age (<50; >=50 to <65; >= 65 years at baseline)
- CDC classification (based on screening information from the parent study)
- Gender
- Race

### 3. SUBJECT INFORMATION

### 3.1. Demographics and Baseline Characteristics

The following parameters will be analyzed:

- Gender (male/female)
- Race (from parent studies)
- Age at baseline
- Age at baseline by categories ( $<50, \ge 50$  to  $<65, \ge 65$ )
- Country/site
- History of Hepatitis B/C
- History of Hepatitis B
- History of Hepatitis C
- Clade

### 3.2. Disposition Information

Discontinuations, plus reasons for discontinuation will be analyzed:

Summary statistics (count, percentage and rate per 100 person-years) will be provided. Rate per 100 person-years is calculated as (the total number of discontinuations x 100) divided by (the

total number of days summed over all subjects)/365.25. Exact 95% confidence intervals<sup>4</sup> for the number of discontinuation per 100 person-years will also be provided.

### 3.3. Extent of Exposure

Exposure is defined as the duration of RPV treatment during the active treatment phase (in Days). The extent of exposure will be summarized in years, and the total person-years-of exposure will be provided.

Treatment duration is calculated as follows: last day of treatment phase - Day of first dose + 1. Note that the above definition implies that drug interruptions are ignored in calculating exposure.

The total person-years-of-exposure will be calculated by taking the sum of the RPV treatment duration (years) over all subjects.

In addition, the proportion of subjects in the study exposed to RPV will be tabulated using 48-week intervals, i.e. based on 1 x 48 weeks (337 days), 2 x 48 weeks (673 days), etc. as cut-points (see Table 2).

#### 3.4. Protocol Deviations

Major protocol deviations will be tabulated and listed.

#### 3.5. Concomitant Medications

Concomitant therapies are defined as therapies listed on the concomitant medications (CM) domain. Concomitant medications are allocated to each phase during which they were administered, based on their start and end dates. For phase allocation, the following rules are applied to deal with (partially) missing start or end dates:

- a start date with the day only missing has the day imputed with the first day of the month;
- a start date with the day and month missing has the day imputed with the 1st of January;
- an entirely missing start date is considered as having started before the study;
- an end date with the day only missing has the day imputed with the last day of the month;
- an end date with the day and month missing has the day imputed with the 31st of December:
- an entirely missing end date is considered as having ended after the study.

Number and percent of subjects per ARV therapy (as started or ongoing at baseline) will be summarized. In addition, all ARV and non-ARV therapies will be listed separately. A separate listing for all subjects who switched ARV therapy during treatment will also be listed. Note: combination drugs will be split into their respective compounds.

### 3.6. Adherence

Treatment adherence is defined based on drug accountability from tablet counts.

The following parameters are derived over the entire treatment period.

#### **Drug accountability**

Amount to be taken = (number of days since start of treatment x number of tablets to be taken per day).

Number of days since start of treatment in C222 is:

- based on <u>last RPV study medication intake date</u> (if available) or, in case subject discontinued and last RPV study medication intake date is missing, <u>discontinuation</u> date
- if not available, the last dispensation visit will be used.

<u>Actual amount taken in C222</u> = (number of tablets dispensed – number of tablets returned)

Tablets dispensed after or on the date of last dose (based on exposure data) should not be taken into account if there is no information on all dispensed tablets available.

<u>Level of adherence</u> = (actual amount taken / amount to be taken) x 100%

Treatment adherence is defined as:

- adherent: the level of adherence is > 95%
- non-adherent: the level of adherence is < 95%

Additionally, following categories of level of adherence will be defined:

- > 95%
- [80%; 95%]
- [65%; 80%]
- [50%; 65%]
- < 50%

The numbers and percentages of subjects adherent during the trial will be tabulated and descriptive statistics of adherence (%) will be shown.

Interruptions (for AEs) are not to be considered for the calculation of adherence, i.e. they will not be subtracted from the amount to be taken.

Results will be summarized for RPV only.

#### 4. EFFICACY

# 4.1. Analysis Specifications

### 4.1.1. Level of Significance

No statistical testing will be done as this is a single arm trial.

### 4.1.2. Data Handling Rules

Viral load testing was performed locally using several assays. Viral load will be analyzed irrespective of which viral load assay was used (there will be no separate reporting). Regardless

of which assay was used to define response (undetectable)/loss of response (detectable) in the analysis, a cut-off of 50 and 200 copies/mL<sup>2</sup> will be applied.

Imputation of left censored values: 49 copies/mL for values below the detection limit.

Reanalyzed samples will not be used in any of the calculations or summary statistics.

Only samples obtained during the treatment phase will be used for the analyses.

# 4.2. Efficacy Endpoints

The following viral load parameters will be analyzed:

- **Time to Virologic rebound** defined as the time to (first) HIV-1 RNA ≥50/200 copies/mL. Following rules apply:
  - Virologic rebound needs to be confirmed at 2 consecutive visits with the following exception: loss of response at the last study visit where no confirmation sample is available will be considered as rebound.
  - The analysis will be censored at the time of discontinuation (discontinuation due to ANY reason).
  - This is the time (in days) calculated from baseline until the failure time point.
     Subjects never losing the acquired response will be censored at the end of the treatment phase.

#### - **Time to Treatment failure** is defined as

- The time to virologic rebound (see above) or discontinuation, whichever comes first
- Subjects who would otherwise had continued will be censored at the end of the treatment phase.
- This is the time (in days) calculated from baseline until the failure time point.
   Subjects never losing the acquired response will be censored at the end of the treatment phase.

### 4.2.1. CD4<sup>+</sup> cell count

Actual CD4<sup>+</sup> cell count and change in CD4<sup>+</sup> cell count (absolute) from baseline up to Week 360 by 24 Week intervals.

Change from baseline in CD4<sup>+</sup> count is defined as CD4<sup>+</sup> at a given timepoint - baseline CD4<sup>+</sup>.

- Subjects who discontinued because RPV became commercially available or rolled over to IFD3004 will be censored at that time.
- Subjects who discontinued for any other reason will have their CD4<sup>+</sup> values after discontinuation imputed with their baseline value (baseline from roll-over study), thus resulting in a 0 change.
- Intermittently missing values will be imputed using a last observation carried forward approach.

# 4.2.2. Analysis Methods

For "time to" parameters, Kaplan Meier estimates and 95% CIs will be calculated. Kaplan-Meier curves will be constructed.

In addition, the cumulative number of events (rebound/treatment failure) and the cumulative number per 100 person-years will be summarized by 24-Week treatment period and for the entire treatment period (Week 360 time point). Rate per 100 person-years is calculated as (the number of failures x 100) divided by (the total number of days summed over all subjects)/(365.25). Exact 95% confidence intervals<sup>4</sup> for the number of events per 100 person-years will also be provided.

For continuous parameters, descriptive statistics (n, mean (se), median, and ranges) per time point and graphical display will be presented.

HIV-1 RNA levels will be listed for all subjects with virologic rebound.

### 5. RESISTANCE DETERMINATIONS

Resistance data will only be analyzed if available for at least 20 subjects. If there are less than 20 subjects, resistance data will be listed. Inclusion of subjects for resistance analysis will solely be based on the availability of post-baseline genotypic data within the treatment phase.

Note: no phenotypic data was collected in this trial.

#### 6. SAFETY

Safety results will be summarized for the Treatment phase only; all safety data (including Follow-up phase) will be included in listings.

#### 6.1. Adverse Events

AE incidence (count, percentage) will be tabulated, overall and by SOC/preferred term.

Overall AE summary tables by preferred term/SOC for serious AEs and pregnancies, AEs leading to discontinuation, AEs at least grade 3, AEs at least grade 4, Grade 3-4 rash, HIV-related AEs and AEs at least possibly related to RPV will be presented throughout the treatment phase only; any AEs in the Follow-up phase will be listed only.

AEs are categorized in different groups of AEs of interest (see Appendix 1).

The different classes of events of interest that will be investigated are the following:

- AEs leading to discontinuation
- Skin events of interest (with subcategories: Rash)
- Neuropsychiatric events of interest (with subcategories: Neurologic events of interest, Psychiatric events of interest). The subcategories are based on System Organ Class.
- Potential QT prolongation-related events
- Hepatic events of interest

## Endocrinology events

Note: the above is based on adverse events of interest analyses in previous Phase 3 studies.

Clinical narratives will be written for: deaths, pregnancies, SAEs at least possibly related to RPV, AEs leading to permanent discontinuation of RPV, grade 3/4 AEs of special interest.

### 6.2. Clinical Laboratory Tests

# 6.2.1. Overall Laboratory Safety

Results from local laboratory testing will be included in the analysis. Lab assessments were only collected for following cases: serious AEs, AEs leading to discontinuation, AEs considered at least possibly related to RPV, grade 3/4 rash.

All laboratory values and pregnancy results collected will be listed. Original units will be reported. All lab values will be used, including those from unscheduled laboratory visits and pregnancy results.

Toxicity grades are determined according to the <u>DAIDS grading list</u> (see protocol). More detailed information will be provided in the DPS.

# **REFERENCES**

- 1. Top HIV Med. 2013;21(1):6-14 2013, International Antiviral Society-USA
- 2. O'Connor J et al 2017 Durability of Viral Suppression with first line anti-retroviral therapy in patients with HIV in the UK: an observational cohort study; Lancet HIV. 2017 Jul; 4(7): e295–e302.
- 3. Bennett DE, Camacho RJ, Otelea D, Kuritzkes DR, Fleury H, et al. 2009 Drug Resistance Mutations for Surveillance of Transmitted HIV-1 Drug-Resistance: 2009 Update. PLoS ONE 4(3): e4724. doi:10.1371/journal.pone.000472
- 4. Ulm K: A simple method to calculate the confidence interval of a standardized mortality ratio (SMR); Am J Epidemiol 1990; 131(2): 373-5.

# **APPENDIX 1: ADVERSE EVENTS OF INTEREST**

| AEDECOD | Category | Subcategory |
|-------------------------------------------|---------------|-------------|
| 17-HYDROXYPROGESTERONE INCREASED | ENDOCRINE | |
| ACTH STIMULATION TEST ABNORMAL | ENDOCRINE | |
| ADRENAL ADENOMA | ENDOCRINE | |
| ADRENOCORTICAL INSUFFICIENCY CHRONIC | ENDOCRINE | |
| AMENORRHOEA | ENDOCRINE | |
| BLOOD ALDOSTERONE DECREASED | ENDOCRINE | |
| BLOOD CORTISOL ABNORMAL | ENDOCRINE | |
| BLOOD CORTISOL DECREASED | ENDOCRINE | |
| BLOOD CORTISOL INCREASED | ENDOCRINE | |
| DEHYDROEPIANDROSTERONE DECREASED | ENDOCRINE | |
| DYSFUNCTIONAL UTERINE BLEEDING | ENDOCRINE | |
| HAIR GROWTH ABNORMAL | ENDOCRINE | |
| HYPERTRICHOSIS | ENDOCRINE | |
| HYPOGONADISM | ENDOCRINE | |
| HYPOTRICHOSIS | ENDOCRINE | |
| MENOMETRORRHAGIA | ENDOCRINE | |
| MENORRHAGIA | ENDOCRINE | |
| MENSTRUAL DISORDER | ENDOCRINE | |
| MENSTRUATION DELAYED | ENDOCRINE | |
| MENSTRUATION IRREGULAR | ENDOCRINE | |
| METRORRHAGIA | ENDOCRINE | |
| OVARIAN CYST | ENDOCRINE | |
| PAROVARIAN CYST | ENDOCRINE | |
| PIGMENTATION DISORDER | ENDOCRINE | |
| POLYMENORRHOEA | ENDOCRINE | |
| POSTURAL ORTHOSTATIC TACHYCARDIA SYNDROME | ENDOCRINE | |
| PROGESTERONE ABNORMAL | ENDOCRINE | |
| PROGESTERONE INCREASED | ENDOCRINE | |
| SKIN DISCOLOURATION | ENDOCRINE | |
| SKIN HYPERPIGMENTATION | ENDOCRINE | |
| SKIN HYPOPIGMENTATION | ENDOCRINE | |
| ACUTE HEPATIC FAILURE | HEPATOBILIARY | |
| ALANINE AMINOTRANSFERASE ABNORMAL | HEPATOBILIARY | |
| ALANINE AMINOTRANSFERASE INCREASED | HEPATOBILIARY | |
| ASPARTATE AMINOTRANSFERASE ABNORMAL | HEPATOBILIARY | |
| ASPARTATE AMINOTRANSFERASE INCREASED | HEPATOBILIARY | |
| BILIRUBIN CONJUGATED INCREASED | HEPATOBILIARY | |
| BILIRUBINURIA | HEPATOBILIARY | |
| BIOPSY LIVER | HEPATOBILIARY | |
| BLOOD ALKALINE PHOSPHATASE INCREASED | HEPATOBILIARY | |
| BLOOD BILIRUBIN INCREASED | HEPATOBILIARY | |
| BLOOD BILIRUBIN UNCONJUGATED INCREASED | HEPATOBILIARY | |

| BLOOD LACTATE DEHYDROGENASE INCREASED | HEPATOBILIARY |
|------------------------------------------------------|---------------|
| CHOLELITHIASIS | HEPATOBILIARY |
| CYTOLYTIC HEPATITIS | HEPATOBILIARY |
| GAMMA-GLUTAMYLTRANSFERASE INCREASED | HEPATOBILIARY |
| HEPATIC CIRRHOSIS | HEPATOBILIARY |
| HEPATIC ENZYME ABNORMAL | HEPATOBILIARY |
| HEPATIC ENZYME INCREASED | HEPATOBILIARY |
| HEPATIC FAILURE | HEPATOBILIARY |
| HEPATIC FUNCTION ABNORMAL | HEPATOBILIARY |
| HEPATIC FUNCTION ABNORMAL NOS | HEPATOBILIARY |
| HEPATIC STEATOSIS | HEPATOBILIARY |
| HEPATITIS | HEPATOBILIARY |
| HEPATITIS ACUTE | HEPATOBILIARY |
| HEPATITIS B | HEPATOBILIARY |
| HEPATITIS C | HEPATOBILIARY |
| HEPATOBILIARY DISEASE | HEPATOBILIARY |
| HEPATOMEGALY | HEPATOBILIARY |
| HEPATOSPLENOMEGALY | HEPATOBILIARY |
| HEPATOSPLENOMEGALY NOS | HEPATOBILIARY |
| HEPATOTOXICITY | HEPATOBILIARY |
| HEPATOTOXICITY NOS | HEPATOBILIARY |
| HYDROCHOLECYSTIS | HEPATOBILIARY |
| HYPERBILIRUBINAEMIA | HEPATOBILIARY |
| HYPERBILIRUBINEMIA | HEPATOBILIARY |
| HYPERTRANSAMINASAEMIA | HEPATOBILIARY |
| JAUNDICE | HEPATOBILIARY |
| JAUNDICE NOS | HEPATOBILIARY |
| LIVER DISORDER | HEPATOBILIARY |
| LIVER FATTY | HEPATOBILIARY |
| LIVER FUNCTION TEST ABNORMAL | HEPATOBILIARY |
| LIVER PALPABLE SUBCOSTAL | HEPATOBILIARY |
| TRANSAMINASES INCREASED | HEPATOBILIARY |
| URINE BILIRUBIN INCREASED | HEPATOBILIARY |
| YELLOW SKIN | HEPATOBILIARY |
| ABNORMAL BEHAVIOUR | NEUROPSYCH |
| ABNORMAL DREAMS | NEUROPSYCH |
| ACUTE PSYCHOSIS | NEUROPSYCH |
| ADJUSTMENT DISORDER | NEUROPSYCH |
| ADJUSTMENT DISORDER NOS | NEUROPSYCH |
| ADJUSTMENT DISORDER WITH ANXIETY | NEUROPSYCH |
| ADJUSTMENT DISORDER WITH DEPRESSED MOOD | NEUROPSYCH |
| ADJUSTMENT DISORDER WITH MIXED ANXIETY AND DEPRESSED | NEOROFSICH |
| MOOD | NEUROPSYCH |
| AFFECT LABILITY | NEUROPSYCH |
| AFFECTIVE DISORDER | NEUROPSYCH |

**AGGRESSION NEUROPSYCH AGITATION NEUROPSYCH AGORAPHOBIA NEUROPSYCH** ALCOHOL ABUSE **NEUROPSYCH** ALCOHOL POISONING **NEUROPSYCH** ALCOHOL WITHDRAWAL SYNDROME **NEUROPSYCH** ALCOHOLISM NFUROPSYCH **AMNESIA NEUROPSYCH ANGER NEUROPSYCH ANHEDONIA NEUROPSYCH ANXIETY NEUROPSYCH** ANXIETY DISORDER **NEUROPSYCH APATHY NEUROPSYCH** ATTENTION DEFICIT/HYPERACTIVITY DISORDER **NEUROPSYCH** AUTONOMIC NERVOUS SYSTEM IMBALANCE **NEUROPSYCH BALANCE DISORDER NEUROPSYCH BALANCE IMPAIRED NEUROPSYCH BALANCE IMPAIRED NOS NEUROPSYCH BIPOLAR DISORDER NEUROPSYCH BIPOLAR I DISORDER NEUROPSYCH BOREDOM NEUROPSYCH BRADYPHRENIA NEUROPSYCH BRUXISM NEUROPSYCH CATATONIA NEUROPSYCH** CLAUSTROPHOBIA **NEUROPSYCH CLUSTER HEADACHE NEUROPSYCH COGNITIVE DISORDER NEUROPSYCH COMPLETED SUICIDE NEUROPSYCH CONCENTRATION IMPAIRED** NFUROPSYCH **CONFUSIONAL STATE NEUROPSYCH CONVERSION DISORDER NEUROPSYCH** COORDINATION ABNORMAL **NEUROPSYCH** CRANIAL NEUROPATHY **NEUROPSYCH DECREASED ACTIVITY NEUROPSYCH** DELIRIUM **NEUROPSYCH DELUSION NEUROPSYCH DEPRESSED LEVEL OF CONSCIOUSNESS NEUROPSYCH** DEPRESSED MOOD **NEUROPSYCH DEPRESSION NEUROPSYCH DEPRESSION AGGRAVATED NEUROPSYCH DEPRESSIVE SYMPTOM NEUROPSYCH** DISORIENTATION **NEUROPSYCH** DISSOCIATION **NEUROPSYCH** DISTRACTIBILITY **NEUROPSYCH DISTURBANCE IN ATTENTION NEUROPSYCH** 

| DIZZINESS | NEUROPSYCH |
|---------------------------------|------------|
| DRUG DEPENDENCE | NEUROPSYCH |
| DYSPHORIA | NEUROPSYCH |
| DYSSOMNIA | NEUROPSYCH |
| DYSTHYMIC DISORDER | NEUROPSYCH |
| EARLY MORNING AWAKENING | NEUROPSYCH |
| EMOTIONAL DISORDER | NEUROPSYCH |
| EMOTIONAL DISTRESS | NEUROPSYCH |
| EUPHORIC MOOD | NEUROPSYCH |
| HALLUCINATION | NEUROPSYCH |
| HALLUCINATION, AUDITORY | NEUROPSYCH |
| HALLUCINATION, VISUAL | NEUROPSYCH |
| HALLUCINATIONS, MIXED | NEUROPSYCH |
| HEAD DISCOMFORT | NEUROPSYCH |
| HEADACHE | NEUROPSYCH |
| HEADACHE NOS AGGRAVATED | NEUROPSYCH |
| HEMICEPHALALGIA | NEUROPSYCH |
| HOMICIDAL IDEATION | NEUROPSYCH |
| HYPERKINESIA | NEUROPSYCH |
| HYPERSOMNIA | NEUROPSYCH |
| HYPOMANIA | NEUROPSYCH |
| INITIAL INSOMNIA | NEUROPSYCH |
| INSOMNIA | NEUROPSYCH |
| INSOMNIA EXACERBATED | NEUROPSYCH |
| IRRITABILITY | NEUROPSYCH |
| LETHARGY | NEUROPSYCH |
| LIBIDO DECREASED | NEUROPSYCH |
| LIBIDO DISORDER | NEUROPSYCH |
| LIBIDO INCREASED | NEUROPSYCH |
| LISTLESS | NEUROPSYCH |
| LOSS OF LIBIDO | NEUROPSYCH |
| MAJOR DEPRESSION | NEUROPSYCH |
| MALE ORGASMIC DISORDER | NEUROPSYCH |
| MANIA | NEUROPSYCH |
| MEMORY IMPAIRMENT | NEUROPSYCH |
| MENTAL DISORDER | NEUROPSYCH |
| MENTAL IMPAIRMENT | NEUROPSYCH |
| MENTAL STATUS CHANGES | NEUROPSYCH |
| MIDDLE INSOMNIA | NEUROPSYCH |
| MONONEUROPATHY | NEUROPSYCH |
| MOOD ALTERED | NEUROPSYCH |
| MOOD SWINGS | NEUROPSYCH |
| NEGATIVE THOUGHTS | NEUROPSYCH |
| NERVOUSNESS | NEUROPSYCH |
| NIGHTMARE | NEUROPSYCH |
| ···-··························· | |

**NIGHTMARES NEUROPSYCH** ORGASM ABNORMAL **NEUROPSYCH** PANIC ATTACK **NEUROPSYCH** PANIC DISORDER **NEUROPSYCH** PARAESTHESIA CIRCUMORAL **NEUROPSYCH PARANOIA NEUROPSYCH** PERSONALITY DISORDER **NEUROPSYCH PHOBIA NEUROPSYCH PHOTOPHOBIA NEUROPSYCH** POOR QUALITY SLEEP **NEUROPSYCH** POST-TRAUMATIC STRESS DISORDER **NEUROPSYCH PSYCHIATRIC INVESTIGATION NEUROPSYCH** PSYCHOGENIC ERECTILE DYSFUNCTION **NEUROPSYCH** PSYCHOLOGICAL FACTOR AFFECTING MEDICAL CONDITION **NEUROPSYCH** PSYCHOMOTOR HYPERACTIVITY **NEUROPSYCH** PSYCHOTIC DISORDER **NEUROPSYCH** PSYCHOTIC DISORDER DUE TO A GENERAL MEDICAL CONDITION **NEUROPSYCH RESTLESS LEGS SYNDROME** NEUROPSYCH RESTLESSNESS **NEUROPSYCH** SEASONAL AFFECTIVE DISORDER **NEUROPSYCH SEDATION NEUROPSYCH** SENSATION OF PRESSURE IN EAR **NEUROPSYCH** SENSE OF OPPRESSION **NEUROPSYCH** SLEEP DISORDER **NEUROPSYCH SLEEP DISORDER NOS NEUROPSYCH** SLEEP PHASE RHYTHM DISTURBANCE **NEUROPSYCH SLUGGISHNESS NEUROPSYCH SOCIAL PHOBIA NEUROPSYCH** SOMATOFORM DISORDER NFUROPSYCH **SOMNOLENCE NEUROPSYCH** SOPOR **NEUROPSYCH STRESS NEUROPSYCH** STRESS SYMPTOMS **NEUROPSYCH** SUBSTANCE ABUSE **NEUROPSYCH** SUICIDAL IDEATION **NEUROPSYCH** SUICIDE ATTEMPT **NEUROPSYCH TENSION NEUROPSYCH UVEITIS NEUROPSYCH VERTIGO NEUROPSYCH VISION BLURRED NEUROPSYCH VISUAL DISTURBANCE NEUROPSYCH CARDIAC ARREST** QT PROLONGING EFF **CARDIAC DEATH** QT PROLONGING EFF **CARDIAC FIBRILLATION** QT PROLONGING EFF CARDIO-RESPIRATORY ARREST QT PROLONGING EFF

| ELECTROCARRIOCRAMA OT INTERVAL ARMORMAN | OT DDOLONGING FEE | |
|---|---|---|
| ELECTROCARDIOGRAM QT INTERVAL ABNORMAL ELECTROCARDIOGRAM QT PROLONGED | QT PROLONGING EFF QT PROLONGING EFF | |
| ELECTROCARDIOGRAM REPOLARISATION ABNORMALITY | QT PROLONGING EFF | |
| ELECTROCARDIOGRAM U-WAVE ABNORMALITY | QT PROLONGING EFF | |
| | • | |
| ELECTROCARDIOGRAM U-WAVE BIPHASIC | QT PROLONGING EFF | |
| LONG QT SYNDROME | QT PROLONGING EFF | |
| LONG QT SYNDROME CONGENITAL | QT PROLONGING EFF | |
| LOSS OF CONSCIOUSNESS | QT PROLONGING EFF | |
| SUDDEN CARDIAC DEATH | QT PROLONGING EFF | |
| SUDDEN DEATH | QT PROLONGING EFF | |
| SYNCOPE | QT PROLONGING EFF | |
| TORSADE DE POINTES | QT PROLONGING EFF | |
| VENTRICULAR ARRHYTHMIA | QT PROLONGING EFF | |
| VENTRICULAR FIBRILLATION | QT PROLONGING EFF | |
| VENTRICULAR FLUTTER | QT PROLONGING EFF | |
| VENTRICULAR TACHYARRHYTHMIA | QT PROLONGING EFF | |
| VENTRICULAR TACHYCARDIA | QT PROLONGING EFF | |
| DERMATITIS CONTACT | SKIN | Dermatitis contact |
| URTICARIA CONTACT | SKIN | Dermatitis contact |
| DERMATITIS | SKIN | Dermatitis/Eczema |
| DERMATITIS ATOPIC | SKIN | Dermatitis/Eczema |
| DERMATITIS EXFOLIATIVE | SKIN | Dermatitis/Eczema |
| DERMATITIS NOS | SKIN | Dermatitis/Eczema |
| ECZEMA | SKIN | Dermatitis/Eczema |
| ECZEMA NUMMULAR | SKIN | Dermatitis/Eczema |
| SEBORRHOEIC DERMATITIS | SKIN | Dermatitis/Eczema |
| SKIN INFLAMATION | SKIN | Dermatitis/Eczema |
| SKIN INFLAMMATION | SKIN | Dermatitis/Eczema |
| SKIN INFLAMMATION NOS | SKIN | Dermatitis/Eczema |
| EYE SWELLING | SKIN | Oedema |
| LARYNGEAL OEDEMA | SKIN | Oedema |
| PHARYNGEAL OEDEMA | SKIN | Oedema |
| BLISTER | SKIN | Other |
| CHLOASMA | SKIN | Other |
| DESQUAMATION | SKIN | Other |
| EOSINOPHILIC PUSTULAR FOLLICULITIS | | Other |
| | SKIN | |
| ERYTHEMA NODOSUM | SKIN | Other |
| INFECTED SKIN ULCER | SKIN | Other |
| LIP BLISTER | SKIN | Other |
| LIP ULCERATION | SKIN | Other |
| NEURODERMATITIS | SKIN | Other |
| PENILE ULCERATION | SKIN | Other |
| PHOTOSENSITIVITY REACTION | SKIN | Other |
| PHOTOSENSITIVITY REACTION NOS | SKIN | Other |
| POLYMORPHIC LIGHT ERUPTION | SKIN | Other |

| SCROTAL ULCER | SKIN | Other |
|---------------------------------------------------|------|-------|
| SEBORRHOEA | SKIN | Other |
| SKIN DESQUAMATION | SKIN | Other |
| SKIN DESQUAMATION NOS | SKIN | Other |
| SKIN EXFOLIATION | SKIN | Other |
| SKIN ULCER | SKIN | Other |
| SKIN ULCERATION | SKIN | Other |
| ANGIONEUROTIC OEDEMA | SKIN | Rash |
| DERMATITIS ALLERGIC | SKIN | Rash |
| DERMATITIS MEDICAMENTOSA | SKIN | Rash |
| DRUG ERUPTION | SKIN | Rash |
| DRUG RASH WITH EOSINOPHILIA AND SYSTEMIC SYMPTOMS | SKIN | Rash |
| ERYTHEMA | SKIN | Rash |
| ERYTHEMA GENERALISED | SKIN | Rash |
| ERYTHEMA INDURATUM | SKIN | Rash |
| ERYTHEMA OF EYELID | SKIN | Rash |
| EXANTHEM | SKIN | Rash |
| EXFOLIATIVE RASH | SKIN | Rash |
| EYELID OEDEMA | SKIN | Rash |
| FACE OEDEMA | SKIN | Rash |
| GENERALISED ERYTHEMA | SKIN | Rash |
| GENITAL ERYTHEMA | SKIN | Rash |
| GENITAL RASH | SKIN | Rash |
| PERIORBITAL OEDEMA | SKIN | Rash |
| PRURIGO | SKIN | Rash |
| PRURITUS | SKIN | Rash |
| RASH | SKIN | Rash |
| RASH ERYTHEMATOUS | SKIN | Rash |
| RASH FOLLICULAR | SKIN | Rash |
| RASH GENERALISED | SKIN | Rash |
| RASH MACULAR | SKIN | Rash |
| RASH MACULO-PAPULAR | SKIN | Rash |
| RASH MORBILLIFORM | SKIN | Rash |
| RASH NOS | SKIN | Rash |
| RASH PAPULAR | SKIN | Rash |
| RASH PRURITIC | SKIN | Rash |
| RASH PUSTULAR | SKIN | Rash |
| RASH SCALY | SKIN | Rash |
| RASH URTICARIA-LIKE | SKIN | Rash |
| SKIN REACTION | SKIN | Rash |
| SKIN TOXICITY | SKIN | Rash |
| SWELLING FACE | SKIN | Rash |
| TOXIC SKIN ERUPTION | SKIN | Rash |
| URTICARIA | SKIN | Rash |
| URTICARIA CHRONIC | SKIN | Rash |

| URTICARIA GENERALISED | SKIN | Rash |
|--------------------------|------|----------------|
| URTICARIA LOCALISED | SKIN | Rash |
| URTICARIA NOS | SKIN | Rash |
| URTICARIA PAPULAR | SKIN | Rash |
| DERMATITIS BULLOUS | SKIN | Rash vesicular |
| ERYTHEMA MULTIFORME | SKIN | Rash vesicular |
| RASH VESICULAR | SKIN | Rash vesicular |
| STEVENS-JOHNSON SYNDROME | SKIN | Rash vesicular |